CLINICAL TRIAL: NCT00123487
Title: A Randomized Two-Arm, Multicenter, Open-Label Phase III Study of BMS-354825 Administered Orally at a Dose of 70 mg Twice Daily or 140 mg Once Daily in Subjects With Chronic Myeloid Leukemia in Accelerated Phase or in Myeloid or Lymphoid Blast Phase or With Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia Who Are Resistant or Intolerant to Imatinib Mesylate (Gleevec)
Brief Title: Advanced Chronic Myelogenous Leukemia (CML) - Follow On: Study of BMS-354825 in Subjects With CML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-035; NCT00331396 (obsolete NCT alias)
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Myeloid Leukemia, Chronic, Accelerated Phase; Leukemia, Lymphoblastic, Acute, Philadelphia-Positive
Keywords: Accelerated Phase Chronic Myeloid Leukemia; Lymphoid Blast Phase Chronic Myeloid Leukemia; Myeloid Blast Phase Chronic Myeloid Leukemia; Philadelphia Positive Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dasatinib Twice a Day (BID) (Experimental): 70 mg dasatinib twice a day (BID)
  Interventions: Drug: dasatinib
- dasatinib Once a Day (QD) (Experimental): 140 mg dasatinib once a day (QD)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Tablets, Oral, 70 mg BID, indefinitely, survival study
  Other Names: Sprycel; BMS-354825
  Arms: dasatinib Once a Day (QD)
Drug: dasatinib — Tablets, Oral, 140 mg QD, indefinitely, survival study
  Other Names: Sprycel; BMS-354825
  Arms: dasatinib Twice a Day (BID)

SUMMARY:
This is a phase III study of BMS-354825 in subjects with chronic myelogenous leukemia in accelerated phase, or in myeloid or lymphoid blast phase or with Philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia who are resistant or intolerant to imatinib mesylate (Gleevec).

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Patients with Philadelphia-Positive (Ph+) (or BCR/ABL+) accelerated phase chronic myeloid leukemia, Ph+ (or BCR/ABL+) blast phase chronic myeloid leukemia, or Ph+ (or BCR/ABL+) acute lymphoblastic leukemia whose disease has primary or acquired hematologic resistance to imatinib mesylate or who are intolerant of imatinib mesylate
* Men and women, 18 years of age or older
* Adequate hepatic function
* Adequate renal function
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month before and at least 3 months after the study in such a manner that the risk of pregnancy is minimized
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 - 2

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* A serious uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy
* Uncontrolled or significant cardiovascular disease
* Medications that increase bleeding risk
* Medications that change heart rhythms
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
* History of significant bleeding disorder unrelated to CML
* Concurrent incurable malignancy other than CML
* Evidence of organ dysfunction or digestive dysfunction that would prevent administration of study therapy
* Prior therapy with BMS-35425
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2005-06; Primary Completion 2006-11 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (115):
- United States (26):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Loma Linda University Cancer Center, Loma Linda, California
  - Ucla Dept. Of Medicine, Los Angeles, California
  - Washington Cancer Institute At Washington Hospital Center, Washington D.C., District of Columbia
  - University Of Miami, Miami, Florida
  - Emory University School Of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - The University Of Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University Of Kentucky, Lexington, Kentucky
  - University Of Maryland, Baltimore, Maryland
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Devetten, Marcel, Omaha, Nebraska
  - The Cancer Center At Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute Of New Jersey, New Brunswick, New Jersey
  - New York Presbyterian Hospital, New York, New York
  - The University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Sci Univ, Portland, Oregon
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Local Institution, Capital Federal, Buenos Aires, Argentina
- Australia (5):
  - Local Institution, St Leonards, New South Wales
  - Local Institution, South Brisbane, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Parkville, Victoria
  - Local Institution, Perth, Western Australia
- Local Institution, Vienna, Austria
- Belgium (5):
  - Local Institution, B-leuven
  - Local Institution, Bruges
  - Local Institution, Brussels
  - Local Institution, Charleroi
  - Local Institution, Yvoir
- Brazil (5):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Campinas, São Paulo
  - Local Institution, Morumbi, São Paulo
  - Local Institution, São Paulo, São Paulo
  - Local Institution, Rio de Janeiro
- Canada (3):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Montreal, Quebec
- Czechia (2):
  - Local Institution, Brno
  - Local Institution, Prague
- Denmark (3):
  - Local Institution, Aarhus C, Denmark
  - Local Institution, Herlev
  - Local Institution, Odense C
- Local Institution, Helsinki, Finland
- France (11):
  - Local Institution, Caen
  - Local Institution, Créteil
  - Local Institution, Grenoble
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (6):
  - Local Institution, Dresden
  - Local Institution, Frankfurt
  - Local Institution, Hamburg
  - Local Institution, Leipzig
  - Local Institution, Mainz
  - Local Institution, Mannheim
- Local Institution, Athens, Greece
- Local Institution, Budapest, Hungary
- Local Institution, Dublin, Ireland
- Local Institution, Ramat Gan, Israel
- Italy (6):
  - Local Institution, Bari
  - Local Institution, Bologna
  - Local Institution, Monza
  - Local Institution, Napoli
  - Local Institution, Orbassano (to)
  - Local Institution, Roma
- Local Institution, Rotterdam, Netherlands
- Local Institution, Trondheim, Norway
- Peru (2):
  - Local Institution, Lima, Lima Province
  - Local Institution, Jesus Maria, Lima region
- Local Institution, Quezon City, Philippines
- Poland (6):
  - Local Institution, Gdansk
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Warsaw
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution, Singapore, Singapore
- South Africa (4):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Groenkloof, Gauteng
  - Local Institution, Parktown, Gauteng
  - Local Institution, Observatory, Western Cape
- South Korea (2):
  - Local Institution, Jeollanam-do
  - Local Institution, Seoul
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Valencia
- Sweden (4):
  - Local Institution, Lund
  - Local Institution, Stockholm
  - Local Institution, Umeå
  - Local Institution, Uppsala
- Local Institution, Basel, Switzerland
- Taiwan (2):
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- Local Institution, Bangkok, Thailand
- United Kingdom (5):
  - Local Institution, London, Greater London
  - Local Institution, Glasgow, Scotland
  - Local Institution, Newcastle, Tyne and Wear
  - Local Institution, Edinburgh
  - Local Institution, Liverpool

REFERENCES:
- [Result] Chu SC, Tang JL, Li CC. Dasatinib in chronic myelogenous leukemia. N Engl J Med. 2006 Sep 7;355(10):1062-3; author reply 1063-4. No abstract available. PMID 16960978
- [Derived] Lilly MB, Ottmann OG, Shah NP, Larson RA, Reiffers JJ, Ehninger G, Muller MC, Charbonnier A, Bullorsky E, Dombret H, Brigid Bradley-Garelik M, Zhu C, Martinelli G. Dasatinib 140 mg once daily versus 70 mg twice daily in patients with Ph-positive acute lymphoblastic leukemia who failed imatinib: Results from a phase 3 study. Am J Hematol. 2010 Mar;85(3):164-70. doi: 10.1002/ajh.21615. PMID 20131302
- [Derived] Kantarjian H, Cortes J, Kim DW, Dorlhiac-Llacer P, Pasquini R, DiPersio J, Muller MC, Radich JP, Khoury HJ, Khoroshko N, Bradley-Garelik MB, Zhu C, Tallman MS. Phase 3 study of dasatinib 140 mg once daily versus 70 mg twice daily in patients with chronic myeloid leukemia in accelerated phase resistant or intolerant to imatinib: 15-month median follow-up. Blood. 2009 Jun 18;113(25):6322-9. doi: 10.1182/blood-2008-11-186817. Epub 2009 Apr 15. PMID 19369231
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started June 2005; recruitment completed March 2006; study ended June 2013 (Year 7) when the study closed and all participants were off study treatment. Those participants who were resistant or intolerant to prior imatinib were enrolled.
Pre-assignment Details: 638 participants were enrolled; 27 were not randomized due to: adverse event (1), death (5), other (5), poor/noncompliance (1), no longer met criteria (13), withdrew consent (2). A total of 611 were randomized to treatment; 609 were treated: 2 randomized but not treated due to death (1) and serious adverse event (1).
Groups:
- Dasatinib 140 mg QD: Dasatinib was administered orally at a dose of 140 mg once a day (QD) until disease progression, drug toxicity, withdrawal of consent, investigator or sponsor decision, pregnancy, or decision to do stem cell transplant.
- Dasatinib 70 mg BID: Dasatinib was administered orally at a dose of 70 mg twice a day (BID) until disease progression, drug toxicity, withdrawal of consent, investigator or sponsor decision, pregnancy, or decision to do stem cell transplant.
Period: Randomized
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Started | 306 | 305
Completed | 305 | 304
Not Completed | 1 | 1
Not completed — Death prior to starting treatment | 0 | 1
Not completed — SAE prior to starting treatment | 1 | 0
Period: Treated With Study Drug
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Started | 304 (1 participant randomized to QD but received BID in error. 304 represents actual QD treatment.) | 305 (1 participant randomized to QD but received BID in error. 305 represents actual BID treatment.)
Completed | 0 | 0
Not Completed | 304 | 305
Not completed — Adverse Event | 23 | 22
Not completed — Disease Progression | 141 | 122
Not completed — Physician Decision | 8 | 9
Not completed — Other | 59 | 58
Not completed — Study Drug Toxicity | 62 | 80
Not completed — Withdrawal by Subject | 11 | 13
Not completed — Unknown (case report form lost) | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Population analyzed. Baseline data are based on what participants were randomized to receive and not what they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID | Total
Number analyzed (Participants) | 306 | 305 | 611
Age, Customized [Number; unit: participants]
  Less than (<) 21 years | 5 | 4 | 9
  21 - 45 years | 101 | 83 | 184
  46 - 65 years | 143 | 143 | 286
  66 - 75 years | 49 | 65 | 114
  Greater than (>) 75 years | 8 | 9 | 17
  Not Reported | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 134 | 267
  Male | 173 | 171 | 344
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 38 | 38 | 76
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 17 | 18 | 35
  White | 235 | 236 | 471
  Other | 13 | 9 | 22
  Unknown or Not reported | 3 | 3 | 6
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: participants] — ECOG PS, a 6-item scale to assess disease progression, daily functioning, and appropriate treatment and prognosis. Scale: 0-5, with 0= Fully active, able to carry on all pre-disease performance without restriction and 5=Death.
  participants
    ECOG PS 0 | 138 | 134 | 272
    ECOG PS 1 | 121 | 109 | 230
    ECOG PS 2 | 40 | 58 | 98
    ECOG PS 3 | 7 | 2 | 9
    Not Reported | 0 | 2 | 2
Imatinib Status [Number; unit: participants] — Failure on prior treatment with imatinib due to either resistance to or intolerance of imatinib. Resistance: no hematologic response after a ≥ 4-week treatment or a ≥ 50% increase in blasts after a 2-week treatment (primary resistance); achieved a hematologic response, no longer met criteria consistently on all assessments over a consecutive 2-week period while receiving an imatinib (acquired resistance); progressed while on treatment. Intolerance: Grade ≥ 3 non-hematologic toxicity or a Grade 4 hematologic toxicity lasting for > 2 weeks leading to discontinuation of therapy or dose decrease.
  participants
    Primary Resistance | 43 | 49 | 92
    Acquired Resistance | 192 | 190 | 382
    Intolerance | 67 | 65 | 132
    Missing | 4 | 1 | 5
Participants by Disease Phase [Number; unit: participants] — Chronic Myelogenous Leukemia (CML) consists of a chronic phase lasting three to six years, followed by transformation to an accelerated phase (AP) and blast phases (myeloid and Lymphoid) of much shorter duration. The Philadelphia chromosome (Ph+) status was documented by cytogenetic analysis or by Fluorescent-In Situ Hybridization (FISH) for the presence of a protein kinase (BCR-ABL) on peripheral blood (PB) cells or bone marrow (BM) samples.
  participants
    Accelerated Phase CML | 158 | 159 | 317
    Blast Phase CML - Myeloid | 75 | 74 | 149
    Blast Phase CML - Lymphoid | 33 | 28 | 61
    Ph+ ALL | 40 | 44 | 84

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Major Hematologic Response (MaHR) With 6 Months of Follow-up From Date of Last Enrollment - Randomized Population
Description: MaHR defined by either complete hematologic response (CHR) or no evidence of leukemia (NEL). CHR defined as: white blood cells (WBC) ≤ upper limit of normal (ULN); absolute neutrophil count (ANC) ≥ 1,000/mm^3; platelets ≥ 100,000/mm^3; no blasts or promyelocytes in peripheral blood (PB); bone marrow (BM) blasts ≤ 5%; <5% myelocytes plus metamyelocytes in PB; basophils in PB < 20%; no extra-medullar involvement (including no hepatomegaly or splenomegaly). NEL defined by same criteria as CHR except that platelets and ANC had to satisfy at least one of the following (note that both lower limits had to be satisfied): platelets ≥ 20,000/mm^3 and < 100,000/mm^3; ANC > 500/mm^3 and <1,000/mm^3. After Year 2, Amendment 3 allowed participants to switch from the BID to the QD dosing schedule. Percentage: number of participants with MaHR/number of randomized participants.
Time Frame: Randomization up to 6 months
Population: Participants were analyzed based on the treatment they were randomized to receive (not what they actually received). 95% exact confidence interval (CI) presented.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
percentage of participants | 48.0 [42.3 to 53.8] | 47.9 [42.1 to 53.6]
Statistical Analysis 1: Comparison: Dasatinib 140 mg QD vs Dasatinib 70 mg BID; Primary endpoint was to be assessed at 6-Months: Assuming a 45% MaHR rate in the 70 mg BID participants, the primary efficacy analysis required a total of 540 participants, approximately 270 in each dosing schedule, giving at least 80% power to deduce non-inferiority of the QD schedule relative to the BID schedule if the lower bound of the 95% CI for the difference in MaHR rates (MaHRRQD - MaHRRBID) is greater than -12%; Test type: Non-Inferiority or Equivalence — Non-inferiority of the QD schedule relative to the BID schedule was claimed if the lower bound of the 95% CI for difference (QD - BD) was ≥ -12%; Percent Difference = 0.2, 95% CI 2-sided [-7.8 to 8.1]

2. Secondary Outcome: Percent of Participants With Major Hematological Response (MaHR) With 2 Years of Follow-up From Date of Last Enrollment - Randomized Population
Description: A MaHR was defined as a participant having either CHR or NEL. CHR was defined as: WBC ≤ ULN; ANC ≥ 1,000/mm^3; - platelets ≥ 100,000/mm^3; - no blasts or promyelocytes in PB; BM blasts ≤ 5%; < 5% myelocytes plus metamyelocytes in PB; basophils in PB < 20%; no extra-medullar involvement (including no hepatomegaly or splenomegaly). NEL defined by the same criteria as CHR except that platelets and ANC had to satisfy at least one of the following (both lower limits had to be satisfied): platelets ≥ 20,000/mm^3 and < 100,000/mm^3; ANC > 500/mm^3 and <1,000/mm^3. After Year 2, Amendment 3 allowed participants to switch from the BID to the QD dosing schedule. Percent: number of participants with MaHR /number of participants randomized.
Time Frame: Randomization up to 2 years
Population: Participants were analyzed based on the treatment they were randomized to receive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
percentage of participants | 50.7 [44.9 to 56.4] | 49.8 [44.1 to 55.6]

3. Secondary Outcome: Percent of Participants With Major Hematologic Response (MaHR) by Disease Group - Randomized Population
Description: MaHR was defined by either complete hematologic response (CHR) or no evidence of leukemia (NEL). CHR defined as: white blood cells (WBC) ≤ upper limit of normal (ULN); absolute neutrophil count (ANC) ≥ 1,000/mm^3; platelets ≥ 100,000/mm^3; no blasts or promyelocytes in peripheral blood (PB); bone marrow (BM) blasts ≤ 5%; <5% myelocytes plus metamyelocytes in PB; basophils in PB < 20%; no extra-medullar involvement (including no hepatomegaly or splenomegaly). NEL defined by same criteria as CHR except that platelets and ANC had to satisfy at least one parameter of the following (note that both lower limits had to be satisfied): platelets ≥ 20,000/mm^3 and < 100,000/mm^3; ANC > 500/mm^3 and <1,000/mm^3. After Year 2, Amendment 3 allowed participants to switch from the BID to the QD dosing schedule.. Percentage: participants with MaHR/randomized participants.
Time Frame: Randomization up to 2 years
Population: Participants were analyzed based on the treatment they were randomized to receive. n=number of participants in disease group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
percentage of participants
  Accelerated Phase (n=158, 159) | 66.5 [58.5 to 73.8] | 67.9 [60.1 to 75.1]
  Myeloid Blast Phase (n=75,74) | 28.0 [18.2 to 39.6] | 28.4 [18.5 to 40.1]
  Lymphoid Blast Phase (n=33,28) | 42.4 [25.5 to 60.8] | 32.1 [15.9 to 52.4]
  Ph+ Acute Lymphoblastic Leukemia (n=40,44) | 37.5 [22.7 to 54.2] | 31.8 [18.6 to 47.6]

4. Secondary Outcome: Median Time to Major Hematologic Response (MaHR) - Randomized Population
Description: A participants' time to MaHR was defined as the time from the first dosing date until criteria are first met for CHR or NEL, whichever occurred first. Non-responders were censored at the maximum of the date of last hematologic or cytogenetic assessment. Median time was measured in months.
Time Frame: Day 1 up to 6 months (time of primary endpoint), 2 years
Population: Participants were analyzed based on the treatment they were randomized to receive.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
Months
  6 Months | 1.9 [1.8 to 1.9] | 1.9 [1.5 to 2.0]
  2 Years | 1.9 [1.8 to 1.9] | 1.9 [1.6 to 2.1]

5. Secondary Outcome: Median Duration of a Major Hematologic Response (MaHR) in Those Participants Who Achieved a MaHR During the Study
Description: MaHR was defined by either CHR or no evidence of leukemia NEL. CHR was defined as: WBC ≤ ULN; ANC ≥ 1,000/mm^3; - platelets ≥ 100,000/mm^3; - no blasts or promyelocytes in PB; BM blasts ≤ 5%; < 5% myelocytes plus metamyelocytes in PB; basophils in PB < 20%; no extra-medullar involvement (including no hepatomegaly or splenomegaly). NEL defined by the same criteria as CHR except that platelets and ANC had to satisfy at least one of the following (note that both lower limits had to be satisfied): platelets ≥ 20,000/mm^3 and < 100,000/mm^3; ANC > 500/mm^3 and <1,000/mm^3. Median duration was measured in months.
Time Frame: Day 1 up to 5 years
Population: Participants who achieved a MaHR during the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 156 | 153
Months | 21.1 [14.4 to 30.7] | 24.7 [19.5 to 35.6]

6. Secondary Outcome: Percent of Participants With Overall Hematologic Response - Randomized Population
Description: Overall Hematologic Response (OHR) was defined as CHR, NEL or minor hematologic response (MiHR). CHR was defined as: WBC ≤ ULN; ANC ≥ 1,000/mm^3; - platelets ≥ 100,000/mm^3; - no blasts or promyelocytes in PB; BM blasts ≤ 5%; < 5% myelocytes plus metamyelocytes in PB; basophils in PB < 20%; no extra-medullar involvement (including no hepatomegaly or splenomegaly). NEL defined by the same criteria as CHR except that platelets and ANC had to satisfy at least one of the following (note that both lower limits had to be satisfied): platelets ≥ 20,000/mm^3 and < 100,000/mm^3; ANC > 500/mm^3 and <1,000/mm^3. MiHR defined as: < 15% blasts in BM and in PB; < 30% blasts + promyelocytes in BM and PB; < 20% basophils in PB; No extra-medullary disease other than spleen and liver. Percentage: participants with OHR/ randomized participants.
Time Frame: Randomization up to 6 Months, 2 Years
Population: Participants were analyzed based on the treatment they were randomized to receive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
percentage of participants
  6 Months | 59.2 [53.4 to 64.7] | 57.4 [51.6 to 63.0]
  2 Years | 60.1 [54.4 to 65.7] | 59.0 [53.3 to 64.6]

7. Secondary Outcome: Number of Participants With Best Confirmed Hematologic Response, Major Hematologic Response (MaHR) and Overall Hematologic Response - Randomized Population
Description: Type of hematologic response: CHR defined as: WBC ≤ ULN; ANC ≥ 1,000/mm^3; - platelets ≥ 100,000/mm^3; - no blasts or promyelocytes in PB; BM blasts ≤ 5%; < 5% myelocytes plus metamyelocytes in PB; basophils in PB < 20%; no extra-medullar involvement (including no hepatomegaly or splenomegaly). NEL defined by the same criteria as CHR except that platelets and ANC had to satisfy at least one of the following (note that both lower limits had to be satisfied): platelets ≥ 20,000/mm^3 and <100,000/mm^3; ANC > 500/mm^3 and <1,000/mm^3. Minor Hematologic Response (MiHR): <15% blasts in BM and in PB; < 30% blasts + promyelocytes in BM and PB; < 20% basophils in PB; No extra-medullary disease other than spleen and liver. Major hematologic response (MaHR ) was CHR or NEL. Overall hematologic response was CHR or NEL or MiHR.
Time Frame: Randomization up to 6 months, 2 years
Population: Participants were analyzed based on the treatment they were randomized to receive.
Measure: Number; unit: participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
participants
  Complete Response, 6 months | 94 | 96
  Complete Response, 2 years | 108 | 110
  No Evidence of Leukemia, 6 months | 53 | 50
  No Evidence of Leukemia, 2 years | 47 | 42
  Minor Response, 6 months | 34 | 29
  Minor Response, 2 years | 29 | 28
  No Response, 6 months | 125 | 130
  No Response, 2 years | 122 | 125
  MaHR, 6 months | 147 | 146
  MaHR, 2 years | 155 | 152
  Overall Response, 6 months | 181 | 175
  Overall Response, 2 years | 184 | 180

8. Secondary Outcome: Percent of Participants With Major Cytogenetic Response (MCyR) - Randomized Population
Description: Cytogenetic assessments were performed only for the first 2 years of study. CyR was based on the number of Ph+ metaphases among cells in metaphase on a BM sample. The criteria for CyR were as follows: Complete cytogenetic response (CCyR): 0% Ph+ cells in metaphase in BM; Partial cytogenetic response (PCyR): 1% to 35% Ph+ cells in metaphase in BM; Minor cytogenetic response: 36% to 65% Ph+ cells in metaphase in BM; Minimal cytogenetic response: 66% to 95% Ph+ cells in metaphase in BM; No cytogenetic response: 96% to 100% Ph+ cells in metaphase in BM; Major cytogenetic response (MCyR) was defined as CCyR or PCyR. Percentage: number of participants with MCyR and denominator is number of randomized participants.
Time Frame: Randomization up to 6 Months, 2 Years
Population: Participants were analyzed based on the treatment they were randomized to receive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
percentage of participants
  6 Months | 36.9 [31.5 to 42.6] | 39.3 [33.8 to 45.1]
  2 Years | 41.5 [35.9 to 47.2] | 41.3 [35.7 to 47.1]

9. Secondary Outcome: Number of Participants With Best Cytogenic Response (CyR) - Randomized Population
Description: Cytogenetic assessments were performed only for the first 2 years of study. CyR was based on the number of Ph+ metaphases among cells in metaphase on a BM sample. The criteria for CyR were as follows: Complete cytogenetic response (CCyR): 0% Ph+ cells in metaphase in BM; Partial cytogenetic response (PCyR): 1% to 35% Ph+ cells in metaphase in BM; Minor cytogenetic response: 36% to 65% Ph+ cells in metaphase in BM; Minimal cytogenetic response: 66% to 95% Ph+ cells in metaphase in BM; No cytogenetic response: 96% to 100% Ph+ cells in metaphase in BM.
Time Frame: Randomization up to 6 Months, 2 Years
Population: Participants were analyzed based on the treatment they were randomized to receive.
Measure: Number; unit: participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
participants
  Complete CyR, 6 months | 89 | 84
  Complete CyR, 2 years | 97 | 98
  Partial CyR, 6 months | 24 | 36
  Partial CyR, 2 years | 30 | 28
  Minor CyR, 6 months | 19 | 18
  Minor CyR, 2 years | 13 | 16
  Minimal CyR, 6 months | 47 | 45
  Minimal CyR, 2 years | 43 | 40
  No response, 6 months | 63 | 56
  No response, 2 years | 60 | 51
  Unable to determine, 6 months | 64 | 66
  Unable to determine, 2 years | 63 | 72

10. Secondary Outcome: Median Progression Free Survival (PFS) - Randomized Population
Description: PFS was defined as: Time from randomization until any of the following: Progression of disease (per investigator), or death. For those with blast phase CML or Ph+ ALL, disease progression was: loss of OHR; no decrease from on-study baseline percent blasts in PB or BM on all assessments over a 4-week period after starting maximum dose; absolute increase of at least 50% in PB blast count over a 2-week period after starting maximum dose. For those with accelerated phase CML: the list above also included: Development of blast phase CML at any time after initiation of therapy and development of extra-medullary sites other than spleen or liver. Participants who neither progressed nor died were censored on the date of their last cytogenetic or hematologic assessment. Median duration was measured in months.
Time Frame: Randomization up to 5 Years
Population: Participants were analyzed based on the treatment they were randomized to receive.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
Months | 7.8 [5.9 to 9.2] | 10.4 [7.4 to 12.1]

11. Secondary Outcome: Median Overall Survival (OS) - Randomized Population
Description: OS was defined as time from randomization until date of death. Participants who had not died or who were lost to follow-up were censored on the last date on which the participant was known to be alive. Median duration was measured in months.
Time Frame: Randomization up to 5 Years
Population: Participants were analyzed based on the treatment they were randomized to receive.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
Months | 17.7 [12.5 to 23.5] | 22.4 [18.0 to 32.1]

12. Secondary Outcome: Progression Free Survival (PFS) and Overall Survival (OS) at 24, 36, 48, and 60 Months - Randomized Population
Description: PFS was defined as time from randomization until any of the following: Progression of disease (per investigator), or death. For those with blast phase CML or Ph+ ALL, disease progression was: loss of OHR; no decrease from on-study baseline percent blasts in PB or BM on all assessments over a 4-week period after starting maximum dose; absolute increase of at least 50% in PB blast count over a 2-week period after starting maximum dose. For those with accelerated phase CML: the list above also included: Development of blast phase CML at any time after initiation of therapy and development of extra-medullary sites other than spleen or liver. Participants who neither progressed nor died were censored on the date of their last cytogenetic or hematologic assessment. OS was defined as time from randomization until date of death. Participants who had not died or were lost to follow-up were censored on the last date they were known to be alive. Median duration was measured in months.
Time Frame: 24 months, 36 months, 48 months, 60 months
Population: Participants were analyzed based on the treatment they were randomized to receive. Kaplan-Meir estimates of PFS or OS (95% Confidence Interval) are provided below.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 306 | 305
percentage of participants
  PFS at 24 Months | 29.5 [24.2 to 34.8] | 33.1 [27.4 to 38.8]
  PFS at 36 Months | 24.1 [19.0 to 29.1] | 26.6 [21.0 to 32.1]
  PFS at 48 Months | 19.8 [15.0 to 24.6] | 20.5 [15.1 to 25.9]
  PFS at 60 Months | 16.9 [12.3 to 21.5] | 15.9 [10.5 to 21.2]
  OS at 24 Months | 43.3 [37.5 to 49.0] | 48.7 [42.9 to 54.5]
  OS at 36 Months | 37.1 [31.4 to 42.8] | 42.5 [36.6 to 48.3]
  OS at 48 Months | 32.7 [27.1 to 38.3] | 38.2 [32.4 to 44.0]
  OS at 60 Months | 28.8 [23.4 to 34.3] | 36.1 [30.3 to 41.8]

13. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation and Drug-related Fluid Retention AEs, up to Year 7 in Treated Participants
Description: With protocol Amendment 6, the duration of the study was extended for 2 additional years (7 years total) for participants who continued to have clinical benefit and no feasible alternate access to dasatinib. However, after Year 5 the requirement to follow participants for survival and to collect other efficacy data was removed from the protocol for the remainder of the study. Only AEs and SAEs were collected up to Year 7. On-study AEs and SAEs were graded by severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. The investigator AE terms were coded and grouped by preferred term and system organ class using the Medical Dictionary for Regulatory Activities (MedDRA), version 16.0.
Time Frame: Day 1 to Year 7
Population: All participants who received at least one dose of study drug were analyzed. Participants were analyzed based on the treatment they actually received, not what they were randomized to receive.
Measure: Number; unit: participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 304 | 305
participants
  Deaths | 203 | 186
  Death within 30 Days | 66 | 63
  SAEs | 228 | 236
  AEs Leading to Discontinuation | 118 | 114
  Drug-related Fluid Retention | 109 | 137

14. Secondary Outcome: Number of Participants With Normal Baseline Versus Worst Grade 3/4 Hematology Laboratory Abnormalities up to Year 2 in Treated Participants
Description: Laboratory abnormalities were graded according to the National Cancer Institute Common Terminology Criteria (NCI CTC) version 3.0. CTC Grade 3 and 4 criteria are defined as follows: White blood cells (WBC): Grade (Gr) 3:<2.0 to 1.0*10^9/L, Gr 4:<1.0*10^9/L. Absolute neutrophil count (ANC): Gr 3:<1.0 to 0.5*10^9/L, Gr 4:<0.5*10^9/L. Platelet count Gr 3:<50.0 to 25.0*10^9/L, Gr 4:<25.0 to 10^9/L. Hemoglobin Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL. Baseline was laboratory value obtained within 2 weeks prior to randomization.
Time Frame: Baseline to Year 2
Population: All participants who received at least one dose of study drug were analyzed. Participants were analyzed based on the treatment they actually received, not what they were randomized to receive. Those participants who did not have a parameter reported at baseline are indicated.
Measure: Number; unit: participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 304 | 305
participants
  WBC | 129 | 114
  WBC not reported at baseline | 2 | 2
  Platelets | 64 | 79
  Platelets not reported at baseline | 2 | 2
  Hemoglobin | 12 | 13
  Hemoglobin not reported at baseline | 2 | 2
  ANC | 127 | 143
  ANC not reported at baseline | 9 | 8

15. Secondary Outcome: Number of Participants With Grade 4 Myelosuppression Determined From Hematology Evaluations
Description: Laboratory abnormalities were graded according to the National Cancer Institute Common Terminology Criteria (NCI CTC) Version 3.0. Grade 4 hematology evaluations used to determine myelosuppression included: WBC: <1.0*10^9/L. ANC: <0.5*10^9/L. Platelet count <25.0 to 10^9/L.
Time Frame: Day 1 up to Year 7
Population: All participants who received at least one dose of study drug and had laboratory evaluations available were analyzed. Participants were analyzed based on the treatment they actually received, not what they were randomized to receive.
Measure: Number; unit: participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 299 | 303
participants
  WBC (n=299, 303) | 64 | 72
  Platelets(n=299, 303) | 167 | 164
  ANC (n=299, 303) | 132 | 142

16. Secondary Outcome: Number of Participants With Normal Baseline Versus Worst Grade 3/4 Biochemistry Laboratory Abnormalities up to Year 2 in Treated Participants
Description: Laboratory abnormalities were graded according to the NCI CTC version 3.0. Grade 3 and 4 criteria were defined as follows: Upper limit of normal (ULN). Alanine transaminase (ALT) Grade (Gr) 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. Aspartate aminotransferase (AST) Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. Total bilirubin Gr 3: >3.0 to 10..0*ULN; Gr 4: >10.0.0*ULN. Serum creatinine (H) Gr 3: >3.0 to 6.0*ULN; Gr 4: >6.0*ULN. Calcium (L) Gr3: 6.0-7.0; Gr 4: <6.0 mg/dL; Phosphorus (L): Gr 3: <2.0 - 1.0 mg/dL , Gr 4: <1.0 mg/dL. Non-hematologic laboratory results were not collected beyond Year 2. Baseline values were obtained within 2 weeks prior to randomization.
Time Frame: Baseline to Year 2
Population: All participants who received at least one dose of study drug were analyzed. Participants were analyzed based on the treatment they actually received, not what they were randomized to receive. Participants who did not have a parameter reported at baseline are indicated.
Measure: Number; unit: participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 304 | 305
participants
  Hypophosphatemia | 28 | 26
  Phosphorus not reported at baseline | 14 | 20
  Hypocalcemia | 14 | 9
  Calcium not reported at baseline | 5 | 13
  Elevated ALT | 8 | 4
  ALT not reported at baseline | 4 | 4
  Elevated AST | 3 | 2
  AST not reported at baseline | 3 | 6
  Elevated Bilirubin | 4 | 3
  Bilirubin not reported at baseline | 2 | 7
  Elevated Serum Creatinine | 4 | 2
  Serum Creatinine not reported at baseline | 1 | 3

17. Secondary Outcome: Number of Participants With Changes From Baseline in QT Interval Corrected With Fridericia Formula (QTcF) up to Year 2 in Treated Participants
Description: A12-lead electrocardiogram (ECG) was obtained at baseline (baseline=within 2 weeks prior to randomization) and once between Days 8 and 29. Additional ECGs were done at the Investigator's discretion. ECGs were read centrally. The QT interval corrected with Fridericia formula is presented with categories of changes from baseline (BL) in milliseconds (msec).
Time Frame: Baseline to Year 2
Population: All participants who received at least one dose of study drug and had appropriate baseline and on-study ECG data available were analyzed. Participants were analyzed based on the treatment they actually received, not what they were randomized to receive.
Measure: Number; unit: participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 269 | 257
participants
  QTcF <-60 msec change from BL | 4 | 7
  -60 - < -30 msec change from BL | 13 | 15
  -30 - < 0 msec change from BL | 88 | 65
  0 - 30 msec change from BL | 114 | 125
  > 30 - 60 msec change from BL | 31 | 24
  > 60 msec change from BL | 19 | 21

18. Secondary Outcome: Number of Participants With Maximal QTcF Intervals up to Year 2 in Treated Participants
Description: A12-lead ECG was obtained at baseline (baseline=within 2 weeks prior to randomization) and once between Day 8 and 29. Additional ECGs were done at the Investigator's discretion. ECGs were read centrally. QT Interval corrected with Fridericia formula was measured in msec.
Time Frame: Baseline up to Year 2
Population: All participants who received at least one dose of study drug and had appropriate ECG data available were analyzed. Participants were analyzed based on the treatment they actually received, not what they were randomized to receive.
Measure: Number; unit: participants
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Number analyzed (Participants) | 280 | 270
participants
  Maximum QTcF Interval < 450 msec | 252 | 239
  Maximum QTcF Interval 450 - 500 msec | 21 | 26
  Maximum QTcF Interval > 500 msec | 7 | 5

ADVERSE EVENTS:
Time Frame: Day 1 up to 7 years
Description: Participants who received at least one dose of study drug were analyzed. Participants were analyzed based on the treatment they actually received, not what they were randomized to receive.
Arm/Group | Dasatinib 140 mg QD | Dasatinib 70 mg BID
Serious Adverse Events (participants affected / at risk) | 228/304 | 236/305
Other Adverse Events (participants affected / at risk) | 289/304 | 290/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib 140 mg QD (N=304) | Dasatinib 70 mg BID (N=305)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Alanine aminotransferase (Investigations) | 1 | 0
Arachnoiditis (Nervous system disorders) | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 3
Biopsy lymph gland (Investigations) | 0 | 1
Blast cell proliferation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 2 | 0
Chills (General disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 1
Cystitis (Infections and infestations) | 3 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 28 | 29
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lung abscess (Infections and infestations) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Pneumonia (Infections and infestations) | 26 | 27
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Quadriparesis (Nervous system disorders) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Systemic mycosis (Infections and infestations) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 8
Central nervous system haemorrhage (Nervous system disorders) | 5 | 3
Chest pain (General disorders) | 0 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 2 | 0
Generalised oedema (General disorders) | 0 | 2
Gingival pain (Gastrointestinal disorders) | 0 | 1
Hernia obstructive (General disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 3
Pseudomembranous colitis (Infections and infestations) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Sciatica (Nervous system disorders) | 1 | 0
Septic shock (Infections and infestations) | 3 | 4
Spinal cord compression (Nervous system disorders) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 3
Staphylococcal infection (Infections and infestations) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 4
Systolic dysfunction (Cardiac disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Troponin T increased (Investigations) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Vasculitis (Vascular disorders) | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 2
Fatigue (General disorders) | 4 | 2
Febrile infection (Infections and infestations) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Infection (Infections and infestations) | 15 | 9
Ischaemia (Vascular disorders) | 0 | 1
Leukaemic infiltration brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 5
Neutrophil count (Investigations) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 1
Pain (General disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Poor venous access (Vascular disorders) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Sepsis (Infections and infestations) | 5 | 15
Sinus bradycardia (Cardiac disorders) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 9
White blood cell count increased (Investigations) | 1 | 2
Abscess oral (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Blast cell count increased (Investigations) | 2 | 3
Blood creatinine (Investigations) | 0 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 2 | 0
Death (General disorders) | 4 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Device related infection (Infections and infestations) | 4 | 3
Diverticulitis (Infections and infestations) | 0 | 2
Erysipelas (Infections and infestations) | 1 | 0
Granulocyte count (Investigations) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 4
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 9 | 8
Oral infection (Infections and infestations) | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 34 | 50
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Pyrexia (General disorders) | 20 | 38
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 8
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 2
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Stupor (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 1
Anal infection (Infections and infestations) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Aspartate aminotransferase (Investigations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 3
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 15
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 1
Haemorrhoid infection (Infections and infestations) | 1 | 1
Headache (Nervous system disorders) | 3 | 8
Hypotension (Vascular disorders) | 4 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 7 | 5
Lobar pneumonia (Infections and infestations) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 3 | 2
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Skin infection (Infections and infestations) | 1 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Streptococcus test positive (Investigations) | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Arrhythmia (Cardiac disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 3
Cellulitis (Infections and infestations) | 5 | 2
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 3
Circulatory collapse (Vascular disorders) | 0 | 1
Colostomy (Surgical and medical procedures) | 1 | 0
Corynebacterium test positive (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Demyelinating polyneuropathy (Nervous system disorders) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 14 | 15
Disease progression (General disorders) | 2 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1
Encephalomalacia (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 | 13
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 1 | 1
Haemoglobin (Investigations) | 3 | 3
Haemorrhage intracranial (Nervous system disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Renal failure (Renal and urinary disorders) | 7 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Sudden death (General disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Aspergillus infection (Infections and infestations) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign intracranial hypertension (Nervous system disorders) | 0 | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Cataract (Eye disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 3
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cytomegalovirus infection (Infections and infestations) | 1 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 1
Effusion (General disorders) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Localised infection (Infections and infestations) | 0 | 1
Monoplegia (Nervous system disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Necrotising panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
No therapeutic response (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 8
Panic attack (Psychiatric disorders) | 0 | 1
Platelet count (Investigations) | 2 | 6
Renal failure acute (Renal and urinary disorders) | 6 | 2
Sinusitis (Infections and infestations) | 2 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 12 | 25
Aphasia (Nervous system disorders) | 1 | 0
Aplasia (Congenital, familial and genetic disorders) | 1 | 0
Asthenia (General disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Blood creatinine increased (Investigations) | 2 | 1
Blood potassium decreased (Investigations) | 0 | 1
Caecitis (Gastrointestinal disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Central nervous system infection (Infections and infestations) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 | 21
Colitis (Gastrointestinal disorders) | 7 | 5
Enteritis (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 4
Haematuria (Renal and urinary disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Labile blood pressure (Vascular disorders) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Leukaemic infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Lung infection (Infections and infestations) | 2 | 4
Motor dysfunction (Nervous system disorders) | 1 | 0
Multi-organ failure (General disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 3 | 5
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Sinusitis aspergillus (Infections and infestations) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 27
Troponin increased (Investigations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 3
Varicella (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib 140 mg QD (N=304) | Dasatinib 70 mg BID (N=305)
Bone pain (Musculoskeletal and connective tissue disorders) | 30 | 25
Chills (General disorders) | 12 | 19
Constipation (Gastrointestinal disorders) | 44 | 37
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 16
Oral herpes (Infections and infestations) | 22 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 48 | 37
Pneumonia (Infections and infestations) | 17 | 17
Abdominal pain upper (Gastrointestinal disorders) | 24 | 17
Chest pain (General disorders) | 35 | 22
Nasopharyngitis (Infections and infestations) | 21 | 18
Pruritus (Skin and subcutaneous tissue disorders) | 29 | 25
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 21
Dizziness (Nervous system disorders) | 26 | 26
Fatigue (General disorders) | 86 | 90
Hypertension (Vascular disorders) | 24 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 33 | 30
Nausea (Gastrointestinal disorders) | 103 | 91
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 33 | 16
Pain (General disorders) | 15 | 18
Vomiting (Gastrointestinal disorders) | 81 | 81
Weight decreased (Investigations) | 51 | 53
Neutropenia (Blood and lymphatic system disorders) | 36 | 35
Night sweats (Skin and subcutaneous tissue disorders) | 19 | 15
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 72 | 106
Pyrexia (General disorders) | 112 | 99
Abdominal pain (Gastrointestinal disorders) | 37 | 39
Decreased appetite (Metabolism and nutrition disorders) | 51 | 65
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 79 | 88
Gingival bleeding (Gastrointestinal disorders) | 16 | 13
Headache (Nervous system disorders) | 112 | 100
Weight increased (Investigations) | 32 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 | 45
Diarrhoea (Gastrointestinal disorders) | 131 | 147
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 31 | 22
Haematoma (Vascular disorders) | 11 | 19
Anxiety (Psychiatric disorders) | 19 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 84 | 93
Dyspepsia (Gastrointestinal disorders) | 24 | 15
Oedema peripheral (General disorders) | 52 | 65
Petechiae (Skin and subcutaneous tissue disorders) | 26 | 21
Anaemia (Blood and lymphatic system disorders) | 33 | 34
Asthenia (General disorders) | 35 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 34
Contusion (Injury, poisoning and procedural complications) | 18 | 8
Depression (Psychiatric disorders) | 19 | 22
Haemorrhoids (Gastrointestinal disorders) | 16 | 16
Insomnia (Psychiatric disorders) | 19 | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 20
Pericardial effusion (Cardiac disorders) | 4 | 19
Rash (Skin and subcutaneous tissue disorders) | 58 | 65
Stomatitis (Gastrointestinal disorders) | 17 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 45 | 40
Upper respiratory tract infection (Infections and infestations) | 31 | 29
Urinary tract infection (Infections and infestations) | 25 | 16

LIMITATIONS AND CAVEATS:
Amendment 3 (7 March 2007) allowed participants to switch from BID to QD dosing. Therefore, results for BID summarized by treatment group after Year 2 may not be a complete reflection of the BID experience and should be interpreted with this in mind.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.